CLINICAL TRIAL: NCT03022487
Title: Multicentre Investigation of Novel Electrocardiogram Risk Markers in Ventricular Arrhythmia Prediction (MINERVA)
Brief Title: Multicentre Investigation of Novel Electrocardiogram Risk Markers in Ventricular Arrhythmia Prediction
Acronym: MINERVA
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0556; 186618 (Other: IRAS Number); 16/NI/0069 (Other: Ethics Reference)
Record Dates: First submitted 2017-01-09; First posted 2017-01-16 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2022-05

CONDITIONS: Ventricular Arrythmia; Ischemic Cardiomyopathy
Keywords: Sudden Cardiac Death (SCD); implantable cardioverter defibrillator; electrophysiological; EP; Ischaemic cardiomyopathy; Ventricular Arrhythmia; ICD
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- ICD Patients with Ischaemic cardiomyopathy: A standard 30-minute electrophysiological (EP) cardiac stimulation protocol will be performed at the end of the ICD implant at baseline. Participants will be followed up for at least 12 months for endpoints.

SUMMARY:
This is a prospective open label single blinded multi-centre observational study involving a study group of patients already undergoing implantable cardioverter-defibrillator (ICD)(including Cardiac resynchronisation therapy device (CRT-D)) implant. A standard 30-minute electrophysiological (EP) cardiac stimulation protocol will be performed at the end of the ICD implant at baseline. This EP test will be performed whilst measuring a 12-lead ECG and will be correlated with event rates to establish their effectiveness in predicting arrhythmia risk. The minimum follow up period should be 18 months and maximum of 3 years, which is how long the study is funded for. This study is not randomised as all study patients will be receiving the EP study performed at baseline. A minimum of 440 patients will be recruited to document event data at standard clinical ICD follow up intervals - equating to a maximum of 6 visits. Blinding will be maintained at the core lab were the ECG analysis will be performed by a nominated researcher who will not have details of patient health status.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Male or Female, aged 18 years or above
* Female participants of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study
* Diagnosed with a history of ischaemic cardiomyopathy
* Stable, as define as no more than a 100% increase or a 50% decrease, dose of current regular medication as standard for patients at risk of ventricular arrhythmia for at least 4 weeks prior to study entry
* Able (in the Investigators opinion) and willing to comply with all study requirements
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study
* Patients must be able to attend follow up at the study site until the study closure
* Attending for first time primary prevention ICD (including CRT-D) implantation under THE National Institute for Health and Care Excellence (NICE) criteria
* Patients must be able to read and understand English
* Stable dose of current regular medication for at least 4 weeks prior to study entry

Exclusion Criteria:

* Within 28 days since acute coronary syndrome/cardiac surgery
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study: for example - awaiting coronary revascularisation
* Female participants who are pregnant, lactating or planning pregnancy during the course of the study
* Contraindications for electrophysiological study

  * Haemodynamic instability
  * Severe valvular heart disease as define by British Society of Echocardiography (BSE) guidelines
  * Symptomatic coronary artery disease (unstable or refractory angina)
  * Stroke within the last 12 months
* Significant renal disease stage i.e. Chronic Kidney Disease stage 5 (requiring renal replacement therapy and / or Estimated glomerular filtration rate (eGFR) <15), or severe liver disease (end stage or presence of cirrhosis)
* Participants who have participated in another research study involving an investigational product in the past 12 weeks
* Undergone ICD implantation where the right ventricular lead is non-apically positioned e.g. positioned septally
* Clinically judged by a cardiologist to require a ventricular tachycardia (VT) therapy zone less than or equal to 200 bpm
* Any other significant disease or disorders which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study. Specific concerns should be discussed with the Chief / Co - Investigators
* Any other interventional research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 440 patients with Ischaemic cardiomyopathy being fitted with an implantable cardioverter-defibrillator (ICDs)
Sampling Method: Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Regional Restitution Instability Index (R2I2), the mean of the standard deviation of the residuals from the mean gradients for each ECG lead across a range of diastolic intervals, will be determined from an EP study carried out at ICD implant. | 12 - 36 months
  * For each lead of the surface ECG, the QTpeak will be plotted as a function of TpeakQ, and gradients were fitted by using 40ms overlapping least squares linear segments as described previously by Taggart et al. [9]. For each lead, in each 40 ms segment, the difference of the gradient from the mean gradient in that 40 ms segment will be calculated. The mean of the standard deviation of these values will be taken as the R2I2.
  * An R2I2 cut-off of 1.03 (no units) will partition the study population into high and low risk groups.
Peak ECG Restitution Slope (PERS), calculated as the peak restitution curve slope taken as a mean across the 12 ECG leads . | 12 - 36 months
  A PERS cut-off of 1.21 (no units) will partition the study population into high and low risk groups.

CONTACTS AND LOCATIONS:
Overall Officials: G. André Ng, Study Chair — University of Leicester
Locations (8):
- United Kingdom (8):
  - Hull and East Yorkshire Hospitals NHS Trust, Cottingham
  - The Dudley Group NHS Foundation Trust, Dudley
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - Barts Health NHS Trust, London
  - Imperial college Healthcare NHS Trust, London
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ng GA, Mistry A, Newton M, Schlindwein FS, Barr C, Bates MG, Caldwell J, Das M, Farooq M, Herring N, Lambiase P, Osman F, Sohal M, Staniforth A, Tayebjee M, Tomlinson D, Whinnett Z, Yue A, Nicolson WB. Rationale and study design of the MINERVA study: Multicentre Investigation of Novel Electrocardiogram Risk markers in Ventricular Arrhythmia prediction-UK multicentre collaboration. BMJ Open. 2022 Jan 3;12(1):e059527. doi: 10.1136/bmjopen-2021-059527. PMID 34980634